CLINICAL TRIAL: NCT03853421
Title: A Double-blind, Placebo-controlled Study in Healthy Volunteers to Determine the Safety and Tolerability of Single, Ascending Subcutaneous Doses of Sevuparin
Brief Title: Placebo-controlled Study to Determine the Safety and Tolerability of Subcutaneous Doses of Sevuparin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Modus Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PKSC01
Record Dates: First submitted 2019-02-15; First posted 2019-02-25 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-02

CONDITIONS: Safety and Tolerability
MeSH Terms: interventions — sevuparin

STUDY DESIGN:
Intervention Model Description: The study will consist of three dose cohorts (3, 6 and 9 mg/kg sevuparin). Subjects in each cohort will receive a single dose of sevuparin or placebo subcutaneously on Day 1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinical study will be performed in a double-blind manner. Only the site pharmacy personnel, who are responsible for preparing the study drug, will have knowledge of the treatment assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose cohort 3 mg/kg sevuparin (Experimental): The study will consist of three dose cohorts (3, 6 and 9 mg/kg sevuparin). Subjects in each cohort will receive a single dose of sevuparin or placebo subcutaneously on Day 1.
  Interventions: Drug: Sevuparin
- Dose cohort 6 mg/kg sevuparin (Experimental): The study will consist of three dose cohorts (3, 6 and 9 mg/kg sevuparin). Subjects in each cohort will receive a single dose of sevuparin or placebo subcutaneously on Day 1.
  Interventions: Drug: Sevuparin
- Dose cohort 9 mg/kg sevuparin (Experimental): The study will consist of three dose cohorts (3, 6 and 9 mg/kg sevuparin). Subjects in each cohort will receive a single dose of sevuparin or placebo subcutaneously on Day 1.
  Interventions: Drug: Sevuparin

INTERVENTIONS:
Drug: Sevuparin — The study will consist of three dose cohorts (3, 6 and 9 mg/kg sevuparin). Subjects in each cohort will receive a single dose of sevuparin or placebo subcutaneously on Day 1.

SUMMARY:
A Double-blind, Placebo-controlled study in Healthy Volunteers to Determine the Safety and Tolerability of Single, Ascending Subcutaneous Doses of Sevuparin

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, sequential cohort, single escalating dose study to explore the safety, tolerability, pharmacokinetics and pharmacodynamics of sevuparin in healthy volunteer adult male and female subjects. The study will consist of three subcutaneous dose cohorts (3, 6 and 9 mg/kg sevuparin). Each dosing cohort will consist of 8 subjects who will be randomized to receive either a single dose of sevuparin or matching placebo in a 3:1 ratio (6 active/2 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form is signed and dated
* Adult male or female subjects, aged ≥18 to ≤65 years of age inclusive;
* Body mass index ≥19.0 to ≤29.0 kg/m2 and a body weight 50.0-100.0 kg
* Subjects must have a negative pregnancy test and subjects of childbearing potential must either be surgically sterile or be willing to practice a highly effective method of contraception
* Subjects must be in good health, as determined by a medical history, physical examination
* Subjects with no clinically significant and relevant history that could affect the conduct of the study.

Exclusion Criteria:

* Recent trauma or injury or history of clinically significant bleeding.
* Clinical evidence of significant or unstable medical illness
* Subjects who have received any prescribed systemic or topical medication
* Subjects who have received aspirin, anti-platelet therapy, anticoagulant therapy and prophylactic and therapeutic LMWH or un-fractioned heparin.
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies)
* Subjects who have received any medications known to chronically alter drug absorption or elimination processes
* Subjects who are still participating in a clinical study
* Subjects who have donated any blood, plasma or platelets
* Subjects with a significant history of drug allergy
* Subjects who have any clinically significant allergic disease
* Subjects who have a supine blood pressure and supine pulse rate higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 40 bpm, respectively
* Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk of participating in the study, such as QTcF interval > 470 ms, or with sinus rhythm with PR interval <110 ms or >210 ms, confirmed by a repeat ECG.
* Screening transaminases (AST, ALT, GGT) ≥ 1.5 times the ULN; estimated glomerular filtration rate (GFR, MDRD equation) < 60 mL/min; APTT above the normal range, INR above 1.4; absolute platelet count <150,000/μL.
* Male subjects who consume more than 3 units of alcohol per day. Female subjects who consume more than 2 units of alcohol per day.
* Subjects with a positive urine drug screen/alcohol test result
* Subjects who smoke more than 6 cigarettes
* Subjects who have positive hepatitis B or hepatitis C antibody or HIV antibodies.
* Subjects who test positive for HIT antibodies at Screening.
* Any relevant condition, behavior, laboratory value or concomitant medication which, in the opinion of the investigator, makes the subject unsuitable for entry into the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of single ascending subcutaneous doses of sevuparin in healthy male and female subjects. | From baseline until day 28
  Number of participants with treatment-related adverse events as assessed by CTCAE

SECONDARY OUTCOMES:
PK characteristics of sevuparin during and after administration of sevuparin as a single subcutanous injection (3 dose co-horts). | Pre dose until day 3
  Maximum Plasma Concentration [Cmax],
PK characteristics of sevuparin during and after administration of sevuparin as a single subcutanous injection (3 dose co-horts). | Pre dose until day 3
  Area Under the Curve [AUC]).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami (CPMI), Miami, Florida, United States